CLINICAL TRIAL: NCT00356967
Title: An International 7-Week, Double-Blind, Placebo-Controlled, 2-Parallel Group Study to Assess the Efficacy of Dianicline 40 mg BID as an Aid to Smoking Cessation in Cigarette Smokers
Brief Title: Efficacy and Safety of Dianicline Versus Placebo as an Aid to Smoking Cessation
Acronym: EURODIAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC5515; EUDRACT : 2006-001009-20
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2008-12-19 (Estimated); Status verified 2008-12

CONDITIONS: Smoking
Keywords: smoking; cessation; tobacco; smoking cessation; tobacco use cessation
MeSH Terms: conditions — Smoking; Smoking Cessation; Tobacco Use Cessation | interventions — dianicline

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: dianicline

SUMMARY:
The primary objective is to demonstrate the efficacy of dianicline as an aid to smoking cessation in cigarette smokers. The main secondary objectives are: to assess the craving for cigarettes, nicotine withdrawal symptoms and the safety of dianicline.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients over the legal age smoking at least 10 cigarettes per day for at least 2 months

Exclusion Criteria:

* Insufficient level of motivation
* Another participant in the household
* Patients with current psychotic disorder or major depressive disorder

The investigator will evaluate whether there are other reasons why a patient may not participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2006-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
to assess the continuous abstinence from tobacco smoking at every visit during the last four weeks of treatment through direct inquiry of patients
exhaled carbon monoxide testing
and plasma cotinine measurements

SECONDARY OUTCOMES:
questionnaire of smoking urge
Hughes and Hatsukami Minnesota Withdrawal Scale to measure nicotine withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (6):
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Hørsholm, Denmark
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Lysaker, Norway
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Bromma, Sweden

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- See also: Related Info — http://www.sanofi-aventis.com